CLINICAL TRIAL: NCT01181102
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy Efficacy and Safety Study of the Oral Factor Xa Inhibitor DU-176b Compared With Enoxaparin Sodium for Prevention of Venous Thromboembolism in Patients After Total Knee Arthroplasty (STARS E-3 Trial)
Brief Title: A Phase 3 Study of DU-176b, Prevention of Venous Thromboembolism in Patients After Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-B-J302
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-02

CONDITIONS: Venous Thromboembolism
Keywords: anticoagulant; venus thromboembolism; thrombosis; thromboembolism; embolism and thrombosis; deep vein thrombosis; DU-176b; Edoxaban; factor Xa; total knee arthroplasty; Enoxaparin sodium
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis; Thromboembolism; Embolism and Thrombosis; Venous Thrombosis | interventions — edoxaban; enoxaparin sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DU-176b (Experimental): DU-176b oral tablets, 30 mg., taken once daily for 2 weeks, initiated within 6 to 24 hours after surgery.
  Interventions: Drug: edoxaban
- enoxaparin sodium (Active Comparator): enoxaparin sodium 20mg (=2000IU) 0.2ml twice daily, subcutaneous injection for 2 weeks, initiated within 24 to 36 hours after surgery.
  Interventions: Drug: enoxaparin sodium

INTERVENTIONS:
Drug: edoxaban
  Arms: DU-176b
Drug: enoxaparin sodium
  Arms: enoxaparin sodium

SUMMARY:
The objective of this study is to assess the efficacy and safety of DU-176b compared with enoxaparin sodium for the prevention of venous thromboembolism in patients after elective total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total knee arthroplasty

Exclusion Criteria:

* Subjects with risks of hemorrhage
* Subjects with thromboembolic risks
* Subjects who weigh less than 40 kg
* Subjects who are pregnant or suspect pregnancy, or subjects who want to become pregnant.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Fuji, Principal Investigator — Osaka Koseinenkin Hospital
Locations (3):
- Japan (2):
  - Osaka
  - Tokyo
- Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Kawai Y, Fuji T, Fujita S, Kimura T, Ibusuki K, Abe K, Tachibana S. Edoxaban versus enoxaparin for the prevention of venous thromboembolism after total knee or hip arthroplasty: pooled analysis of coagulation biomarkers and primary efficacy and safety endpoints from two phase 3 trials. Thromb J. 2016 Dec 1;14:48. doi: 10.1186/s12959-016-0121-1. eCollection 2016. PMID 27980462
- [Derived] Fuji T, Fujita S, Kimura T, Ibusuki K, Abe K, Tachibana S, Nakamura M. Clinical benefit of graduated compression stockings for prevention of venous thromboembolism after total knee arthroplasty: post hoc analysis of a phase 3 clinical study of edoxaban. Thromb J. 2016 Jun 8;14:13. doi: 10.1186/s12959-016-0087-z. eCollection 2016. PMID 27284271
- [Derived] Fuji T, Wang CJ, Fujita S, Kawai Y, Nakamura M, Kimura T, Ibusuki K, Ushida H, Abe K, Tachibana S. Safety and efficacy of edoxaban, an oral factor Xa inhibitor, versus enoxaparin for thromboprophylaxis after total knee arthroplasty: the STARS E-3 trial. Thromb Res. 2014 Dec;134(6):1198-204. doi: 10.1016/j.thromres.2014.09.011. Epub 2014 Sep 21. PMID 25294589

RESULTS

PARTICIPANT FLOW:
Groups:
- DU-176b: DU-176b oral tablets, 30 mg., taken once daily for 2 weeks
  edoxaban
- Enoxaparin Sodium: enoxaparin sodium 20mg(=2000IU)/0.2ml twice daily, subcutaneous injection for 2 weeks
  enoxaparin sodium
Period: Overall Study
Arm/Group | DU-176b | Enoxaparin Sodium
Started | 360 | 356
Safety Analysis Set | 354 | 349
Efficacy Analysis Population | 299 | 295
Completed | 309 | 310
Not Completed | 51 | 46
Not completed — Adverse Event | 28 | 26
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 5 | 6
Not completed — Withdrawal by Subject | 10 | 12

BASELINE CHARACTERISTICS:
Population: Number of baseline participants reflects the efficacy analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | DU-176b | Enoxaparin Sodium | Total
Number analyzed (Participants) | 299 | 295 | 594
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (7.5) | 72.1 (7.8) | 72.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 229 | 474
  Male | 54 | 66 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 299 | 295 | 594
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 26 | 25 | 51
  Japan | 273 | 270 | 543

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Subjects With Venous Thromboembolism Events.
Description: The primary efficacy endpoint was the proportion of subjects who experienced at least one of the thromboembolic events listed below during the period from the start of study treatment to the venography at the end of study treatment.
  * Lower extremity Deep Vein Thrombosis (DVT) confirmed by unilateral venography at the end of study treatment
  * Definite diagnosis of symptomatic Pulmonary Embolism (PE)
  * Symptomatic DVT confirmed before the venography at the end of study treatment The objectives were to verify the non-inferiority of edoxaban to enoxaparin with regard to prevention of venous Thromboembolism (VTE)
Time Frame: 2 weeks
Population: Efficacy Analysis population. 22 (7.4%) - DU-176b 41 (13.9%) - enoxaparin
Measure: Number (95% Confidence Interval); unit: percent of participants with VTE events
Arm/Group | DU-176b | Enoxaparin Sodium
Number analyzed (Participants) | 299 | 295
percent of participants with VTE events | 7.4 [4.4 to 10.3] | 13.9 [10.0 to 17.8]
Statistical Analysis 1: Comparison: DU-176b vs Enoxaparin Sodium; The incidence proportion of thromboembolic events in the DU-176b group (P˅DU) = The incidence proportion of thromboembolic events in the enoxaparin group (P˅E) + Δ (5%). Alternative hypothesis H˅11: P˅DU < P˅E + Δ (level of significance, 0.025; one-sided). If the null hypothesis H˅01 was rejected, the following analysis had to be sequentially performed using the χ2 test statistic. Null hypothesis H˅02: P˅DU = P˅E Alternative hypothesis H˅12: P˅DU ≠ P˅E (level of significance, 0.05; two-sided); Test type: Non-Inferiority or Equivalence — (non-inferiority) When analyzed using the Z test at a one-sided 0.025 significance level, with the addition of a non-inferiority margin of 5% to the incidence in the enoxaparin group. (superiority) The incidence of thromboembolic events for the FAS was compared using the χ2 test (two-sided significance level: 0.05); p < 0.001, non-inferiority:Z test. superiority:χ2 t — non-inferiority:P < 0.001 superiority:P = 0.010; Cox Proportional Hazard = -6.5, 95% CI 2-sided [-11.5 to -1.6]

2. Secondary Outcome: Incidence of Major Bleeding or Clinically Relevant Non-major Bleeding.
Time Frame: 2 weeks
Population: The Safety Analysis Set was defined as all subjects who were enrolled in the study, but excluded those who had significant GCP violations, who did not receive any doses of the study drug, or who had no safety data after the start of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | DU-176b | Enoxaparin Sodium
Number analyzed (Participants) | 354 | 349
percentage of subjects with bleeds | 6.2 [4.1 to 9.2] | 3.7 [2.2 to 6.3]
Statistical Analysis 1: Comparison: DU-176b vs Enoxaparin Sodium; Test type: Superiority or Other; χ2 test = 2.5, 95% CI 2-sided [-0.8 to 5.9]

ADVERSE EVENTS:
Description: The Safety Analysis Set was defined as all subjects who were enrolled in the study, but excluded those who had significant GCP violations, who did not receive any doses of the study drug, or who had no safety data after the start of study treatment.
Arm/Group | DU-176b | Enoxaparin Sodium
Serious Adverse Events (participants affected / at risk) | 10/354 | 11/349
Other Adverse Events (participants affected / at risk) | 237/354 | 256/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b (N=354) | Enoxaparin Sodium (N=349)
postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
stitch abcess (Infections and infestations) | 1 (1) | 0 (0)
carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
convulsion (Nervous system disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b (N=354) | Enoxaparin Sodium (N=349)
wound haemorrhage (Vascular disorders) | 18 (19) | 10 (10)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 22 (25) | 28 (30)
Alanine aminotransferase increased (Investigations) | 25 (25) | 94 (94)
Aspartate aminotransferase increased (Investigations) | 12 (12) | 87 (87)
Gamma-glutamyltransferase increased (Investigations) | 33 (33) | 64 (65)
blood urine present (Investigations) | 34 (35) | 31 (32)
Cystitis (Infections and infestations) | 8 (8) | 6 (6)
Nasopharyngitis (Infections and infestations) | 16 (16) | 15 (15)
rash (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 10 (12)
Vomiting (Gastrointestinal disorders) | 9 (9) | 7 (7)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Blood bilirubin increased (Investigations) | 14 (14) | 7 (8)
Blood lactate dehydrogenase increased (Investigations) | 6 (6) | 16 (16)
Blood triglycerides increased (Investigations) | 9 (9) | 6 (6)
Haemoglobin decreased (Investigations) | 34 (35) | 31 (32)
Blood alkaline phosphatase increased (Investigations) | 34 (35) | 31 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.